CLINICAL TRIAL: NCT06415942
Title: Single Arm Clinical Trial of a Novel Smartphone-based Somatic and Psychological Symptom Monitoring and Decision Support Tool for African American and Spanish Speaking Patients in the Near Postpartum Period
Brief Title: Assessing the Maternal Outcome Monitoring Systems
Acronym: MOMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAU9647; 5R00MD015781-04 (NIH)
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Maternal Death; Maternal Complication of Pregnancy
Keywords: pregnancy related death; patient reported outcomes; mHealth; patient activation
MeSH Terms: conditions — Maternal Death; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MOMS intervention (Experimental): Participants in this condition will receive the MOMS symptom monitoring and decision support intervention. This is a single arm trial.
  Interventions: Other: Maternal Outcome Monitoring and Support system

INTERVENTIONS:
Other: Maternal Outcome Monitoring and Support system — The Maternal Outcome Monitoring and Support system is a mobile health application that allows participants to choose symptoms they may be having that are warning signs of pregnancy related death. They then receive decision support about when they should seek medical care (call their provider or go to an emergency room).

SUMMARY:
Pregnancy-related death is a growing public health issues, which are of particular concern to minority groups, including African-Americans and Spanish-speaking Latinas. Our proposal aims to improve a patient's ability to detect warning signs of pregnancy related death and seek medical care.

DETAILED DESCRIPTION:
Pregnancy-related death (PRD) rates have risen 120-200% in the United States in the past two decades, and experts estimate that 40-60% of these cases are preventable. Improvement initiatives are predominantly hospital-based and rely on perinatal people recognizing their own symptoms and seeking care without ample support or education. We hypothesize that we can improve patients' self-efficacy and decision-making about when to seek care by helping them to self-monitor symptoms and by providing decision support. We propose to develop a mHealth-based, patient-reported outcome (PRO) and decision-support system to help mothers determine when to seek care for warning signs of PRD. Our project focuses on diverse populations facing postpartum disparities, particularly African- American and Spanish-speaking Latina women. This protocol involves a single-arm pilot trial assessing the feasibility and preliminary effectiveness of MOMS/MAMA for improving knowledge and patient activation among postpartum patients.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 28 weeks pregnant
* Receiving healthcare in the United States
* Age 18 years or older
* [Identify as Black or African American race AND able to speak and read English, AND preferred language of English] OR [Identify as Hispanic/Latino Ethnicity AND Spanish able to speak and read Spanish AND preferred language of Spanish]
* Planned delivery at the following NewYork-Presbyterian hospitals: Children's Hospital of New York, Allen Hospital, Weill Cornell Medical Center, Lower Manhattan Hospital

Exclusion Criteria:

* Severe cognitive impairment
* Major psychiatric illness
* Concomitant terminal illness that would preclude participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Patient activation | Baseline to 6 weeks postpartum
  Change in patient activation measured using the validated Patient Activation Measure (PAM)

SECONDARY OUTCOMES:
Knowledge of pregnancy related death warning signs | Baseline to 6 weeks postpartum
  Change in knowledge of warning signs for pregnancy related death

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NewYork-Presbyterian Columbia University Irving Medical Center, New York, New York
  - NewYork-Prebyterian/Weill Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
Data will be shared in the aggregate. There is no plan to make IDP available to other researchers.